CLINICAL TRIAL: NCT07032415
Title: The Effect of a Nutrition Habit Change Program on Lifestyle and Cognitive Function Level in Morbidly Obese Patients
Brief Title: The Effect of Cognitive Function Level in Morbidly Obese Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Principal Investigator, Adem Yüksel, Associate Prof., Kocaeli City Hospital
Other Study IDs: 2025-76
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Obesity; Morbid Obesity
Keywords: bariatric surgery; cognition
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Morbidly Obese Patients

SUMMARY:
Obesity is a disease caused by many factors, such as lifestyle, eating habits, lack of physical activity, hormonal and genetic influences. These different factors make treatment planning difficult. Common treatments include changes in diet and lifestyle, medications, endoscopic methods (like balloon or botox), and surgery. No matter which method is used, the main goal is to help patients lose weight by creating a negative energy balance. To keep the weight off, patients need to maintain a balanced lifestyle in the long term.

However, many treatments are not successful over time. One important part of long-term success is helping patients change their lifestyle and eating habits. A person's cognitive function may affect how they understand and follow these changes. Some studies show that a high body mass index (BMI) is linked to problems with thinking and memory. While weight loss may help improve brain function, the investigators don't yet know how early cognitive differences affect treatment results.

At the obesity center in our hospital, morbidly obese patients receive support from a team of doctors, dietitians, psychologists, and physiotherapists. For at least three months, they attend individual and group sessions to help change their lifestyle and eating habits. This study aims to see how patients' cognitive function affects how much weight they lose by the end of the program.

ELIGIBILITY:
Inclusion Criteria:

* Applying Kocaeli City Hospital's Obesity Center
* Morbid Obesity
* Completing the program

Exclusion Criteria:

* People with psychiatric and neurological diseases
* People using drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbidly obese patients who are added to the Obesity Center and agree to participate in the study are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2025-07-22 (Estimated); Primary Completion 2026-09-10 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Change of Body Mass Index After Nutrition Habit Change Program | 3 months
  Patients weight and height will be used for Body Mass Index calculations

SECONDARY OUTCOMES:
Cognitive Function Change After Nutrition Habit Change Program | 3 months
  MoCA test will be used

CONTACTS AND LOCATIONS:
Overall Officials: Adem Yüksel, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, İzmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No